CLINICAL TRIAL: NCT07002944
Title: Role of Pulsed Radiofrequency of Shoulder Individual Nerves Versus Brachial Plexus in Management of Chronic Post Mastectomy Shoulder Pain: A Prospective Randomized Controlled Study
Brief Title: Pulsed Radiofrequency of Shoulder Individual Nerves Versus Brachial Plexus in Management of Chronic Post Mastectomy Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmina Sayed, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management Department, National Cancer Institute, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP2412-201-087-194
Record Dates: First submitted 2025-05-24; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Pulsed Radiofrequency; Shoulder Individual Nerves Brachial Plexus; Chronic; Post Mastectomy; Shoulder Pain
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Shoulder Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brachial plexus pulsed radiofrequency group (Other): Patients will receive pulsed radiofrequency of brachial plexus with steroids injection.
  Interventions: Other: Brachial plexus pulsed radiofrequency
- Sholder individual nerves pulsed radiofrequency group (Other): Patients will receive shoulder individual nerves pulsed radiofrequency with steroids injection.
  Interventions: Other: Sholder individual nerves pulsed radiofrequency
- Control group (Active Comparator): Patients will receive conservative treatment (paracetamol 1000 tid and pregabalin 75 mg bid; can be increased to 150 mg bid , oxycodone 10 mg oral every 12 hrs .
  Interventions: Other: Control

INTERVENTIONS:
Other: Brachial plexus pulsed radiofrequency — Patients will receive pulsed radiofrequency of brachial plexus with steroids injection.
  Arms: Brachial plexus pulsed radiofrequency group
Other: Sholder individual nerves pulsed radiofrequency — Patients will receive shoulder individual nerves pulsed radiofrequency with steroids injection.
  Arms: Sholder individual nerves pulsed radiofrequency group
Other: Control — Patients will receive conservative treatment (paracetamol 1000 tid and pregabalin 75 mg bid; can be increased to 150 mg bid , oxycodone 10 mg oral every 12 hrs .
  Other Names: Paracetamol +pregabalin +oxycodone
  Arms: Control group

SUMMARY:
this study aims to assess the role of pulsed radiofrequency of the brachial plexus or pulsed radiofrequency of shoulder individual nerves in the management of post-mastectomy shoulder pain.

DETAILED DESCRIPTION:
Breast cancer is the second most common cancer world-wide following lung cancer. It afflicts about 1.7 million patients annually, of which 60% mandate surgery of the breast and/or the axilla, and nearly 20-50% of them may develop post-mastectomy pain syndrome.

Regarding pulsed RF of the brachial plexus, it is not tried up till now for shoulder pain. Since C 5,6,7 are derived from upper and middle trunks of brachial plexus, then innervation of shoulder joint can be blocked by interscalene brachial plexus block or pulsed radiofrequency . Review of literature demonstrated efficacy of PRF of brachial plexus in case studies for other conditions e.g. pain associated with a tumor involving the brachial plexus , refractory stump pain , chemotherapy-induced peripheral neuropathy of the upper limb and radiation-induced brachial plexopathy .

ELIGIBILITY:
Inclusion Criteria:

* Age (18-65) Years.
* American Society of Anesthesiologists (ASA) physical status (II- III).
* Patients with post mastectomy shoulder pain.
* Body mass index (BMI): (20-40) kg/m2.
* Patients on maximum daily dose tramadol ( 450mg ) and still in pain

Exclusion Criteria:

* Patient refusal.
* Known sensitivity or contraindication to drugs used in the study.
* Pregnancy.
* Recent myocardial infarction.
* Hemodynamically unstable.
* Local and systemic sepsis.
* Psychiatric illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in visual Analogue Scale (VAS ) | 24 weeks post postoperatively
  Changes in visual Analogue Scale (VAS )for assessment of pain relief. A 100 mm horizontal line version will be used with 2 ends (left-end means no pain and right-end means the worst pain). This version is preferred in research studies for chronic pain status.

SECONDARY OUTCOMES:
Functional improvement | 24 weeks post postoperatively
  This is a self-reported analysis for the primary outcome after performing pain interventions. It is divided into 4 categories (0-25%) ≈ no or minimal functional improvement, (> 25- 50%) ≈ mild improvement, (> 50-75%) ≈ moderate improvement, and (>75-100%) ≈ marked improvement.
Analgesic consumption | 24 weeks post postoperatively
  Analgesic consumption will be recorded
Patient satisfaction | 24 weeks post postoperatively
  Satisfaction scores of 0 dissatisfied and 10 very satisfied will be assessed
The impact of treatment on the quality of life of the patient | 24 weeks post postoperatively
  The impact of treatment on the quality of life of the patient, which will be assessed by the SF-36 questionnaire.
Incidence of complications | 24 weeks post postoperatively
  Incidence of complications will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author